CLINICAL TRIAL: NCT05372666
Title: Study of the Glycaemic Index of Breads Made From Flour Naturally Rich in Fibre in Healthy Volunteers
Brief Title: Glycaemic Index of Fibre-rich Flours in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulic Meunerie SA (Industry)
Collaborators: Institut Polytechnique UniLaSalle (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Qualista-IG
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Latin square randomization for test products following reference treatment (as per standard protocol)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control IG100 (Placebo Comparator): 1 small bread loaf using T55 standard white flour for a final content of 50 g equivalent digestible carbohydrates
  Interventions: Other: Standard white bread
- Reference WB (Experimental): 1 small bread loaf using T55 Qualista white flour for a final content of 50 g equivalent digestible carbohydrates
  Interventions: Other: Experimental white bread
- Reference HFB (Active Comparator): 1 small bread loaf using T55 standard white flour supplemented with 11 % standard wheat bran (6% dietary fiber content) for a final content of 50 g equivalent digestible carbohydrates
  Interventions: Other: Standard High-fiber bread
- Qualista HFB 01 (Experimental): 1 small bread loaf using T55 Qualista white flour supplemented with 13 % untreated Qualista wheat bran (6% dietary fiber content) for a final content of 50 g equivalent digestible carbohydrates
  Interventions: Other: Experimental High-fiber bread
- Qualista HFB 02 (Experimental): 1 small bread loaf using T55 Qualista white flour supplemented with 13 % pretreated Qualista wheat bran (treatment A - 6% dietary fiber content) for a final content of 50 g equivalent digestible carbohydrates
  Interventions: Other: Experimental High-fiber bread
- Qualista HFB 03 (Experimental): 1 small bread loaf using T55 Qualista white flour supplemented with 13 % pretreated Qualista wheat bran (treatment B - 6% dietary fiber content) for a final content of 50 g equivalent digestible carbohydrates
  Interventions: Other: Experimental High-fiber bread
- Qualista HFB 04 (Experimental): 1 small bread loaf using T55 Qualista white flour supplemented with 13 % pretreated Qualista wheat bran (treatment C - 6% dietary fiber content) for a final content of 50 g equivalent digestible carbohydrates
  Interventions: Other: Experimental High-fiber bread

INTERVENTIONS:
Other: Standard white bread — Bread to be consumed within 10 minutes after 10h fasting
  Arms: Control IG100
Other: Experimental white bread — Bread to be consumed within 10 minutes after 10h fasting
  Arms: Reference WB
Other: Standard High-fiber bread — Bread to be consumed within 10 minutes after 10h fasting
  Arms: Reference HFB
Other: Experimental High-fiber bread — Bread to be consumed within 10 minutes after 10h fasting
  Arms: Qualista HFB 01; Qualista HFB 02; Qualista HFB 03; Qualista HFB 04

SUMMARY:
The project aims to evaluate the glycaemic index of breads from different types of flour. In particular, we aim to understand the glycaemic and insulin responses as well as satiety and sensory profiles of the products.

ELIGIBILITY:
Inclusion Criteria:

* Having a Body Mass Index (BMI) between 18.5 and 30 kg/m²
* Non-smoker for more than three months
* Having signed the informed consent form
* Likely to follow the constraints generated by the study (one morning per week for 9 weeks)
* Social insurance

Exclusion Criteria:

* Pregnant woman
* Subject with a known progressive somatic or psychiatric disease
* Fasting blood glucose greater than 6.1 mmol/L (1.10 g/L), postprandial blood glucose greater than 7.7 mmol/L (1.4 g/L) or known diabetes treated or untreated
* Hyperinsulinemia or a history of insulinoma
* HbA1c greater than 7 %
* History of hypercholesterolemia, hypertension, diabetes or glucose intolerance
* History of food allergy or digestive pathology likely to affect digestion or absorption
* Renal failure
* ASAT or ALAT elevation beyond 1.5 times the upper limit
* Subject consuming more than three glasses per day of alcohol or suffering from various addictions
* Weight change of more than 3 kg in the last three months
* Person participating in another clinical study, or in a period of exclusion from another study
* Person deprived of liberty or under judicial protection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Glycaemic index | glycemia measured over 120 minutes
  percentage area under the curve compared to standard white bread as 100% reference

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche clinique - Centre Hospitalo Universitaire, Amiens, France

IPD SHARING:
Plan to Share IPD: Undecided